CLINICAL TRIAL: NCT06819514
Title: A Phase 1/2, Multicenter, Open-label,Dose-escalation Study to Evaluate the Safety and Efficacy of Intravenous EXG110 in Patients With Fabry Disease
Brief Title: The Safety and Efficacy of Intravenous EXG110 in Patients With Fabry Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXG110-111
Record Dates: First submitted 2025-01-22; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose arm (Experimental): EXG110 injection, use once by intravenous
  Interventions: Drug: EXG110 Injection
- High dose arm (Experimental): EXG110 injection, use once by intravenous
  Interventions: Drug: EXG110 Injection

INTERVENTIONS:
Drug: EXG110 Injection — EXG110 Injection is gene therapy for Fabry Disease , uses a proprietary AAV capsid with improved liver and muscle specificity.

SUMMARY:
A phase 1/2, multicenter, open-label, Dose-escalation study to evaluate the safety and efficacy of intravenous EXG110 in patients with Fabry disease

DETAILED DESCRIPTION:
Phase 1: Dose -escalation，2 Groups Phase 2: Dose- expansion，1 Group

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female
2. Clinical symptoms (at least one Fabry disease related symptom) and genetic diagnosis of Fabry disease
3. Prior or no prior ERT treatment
4. Have renal or cardiac involvement
5. The participant voluntarily participate and are fully informed, fully understood the study, can comply with the requirements of the protocol, and voluntarily provide biological samples for testing according to the requirements of the protocol

Exclusion Criteria:

1. Screening period laboratory test results: a) aspartate aminotransferase or alanine aminotransferase > 1.5× upper limit of normal (ULN);b) Total bilirubin > 1.5× upper limit of normal (ULN);c) Alkaline phosphatase > 2× upper limit of normal (ULN);d) Hypoalbuminemia ≥ grade 2
2. Serum virology test: a) Hepatitis B: Hepatitis B virus surface antigen (HBsAg) positive, and hepatitis B virus-deoxyribonucleic acid (HBV-DNA) higher than the upper limit of normal detection;b) Hepatitis C: if the hepatitis C virus (HCV) antibody is positive, and the hepatitis C virus-ribonucleic acid (HCV-RNA) is higher than the upper limit of normal test value;c) Syphilis: positive for syphilis screening (Tp-Ab) and positive for syphile-specific antibodies;d) HIV: Known human immunodeficiency virus (HIV) positive history or HIV screening positive
3. Current or have a history of serious cardiovascular disease and surgical history
4. Current underlying liver disease or history of liver disease, as assessed by the investigator, that may affect the safety assessment of the product
5. Acute/chronic infection or other chronic disease that the investigator evaluated will increase the risk of participants in the study
6. Those who have a history of epilepsy, mental illness (such as schizophrenia, depression, mania or anxiety, etc.) or obvious mental disorders, and are incapacitated or cognitively incapacitated due to other reasons.
7. Participant with a history of malignant tumor or currently suffering from any malignant tumor (except for the following tumor diseases: skin basal cell carcinoma, cervical carcinoma in situ, breast carcinoma in situ , skin squamous cell carcinoma has been controlled after treatment);
8. Participant with active autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, immune vasculitis, inflammatory bowel disease, etc.);
9. known history of allergy to the components of the investigational products
10. Participant with a history of drug use or drug abuse or alcoholism
11. Has received, or currently receiving, a clinical trial of another investigational drug/medical device or treatment (other than vitamins and minerals) within 3 months prior to signing the informed consent form (or within 5 half-lives of the investigational drug, whichever is longer)
12. Previous treatment with gene therapy products
13. Those who had received live attenuated vaccine/vaccine within 12 weeks prior to screening or planned to receive it during the study
14. Other clinical conditions that the investigators evaluated needed to be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1: To evaluate the safety and tolerability of EXG110 following a single intravenous infusion | 52 weeks
  Adverse events (AEs), serious adverse events (SAEs), dose-limited toxicity types, severity, incidence,
Phase 2: The changes from the baseline of kidney function | 6 months
  Proportion of participants with a reduction in Gb3 inclusion body accumulation to scores 0 (the minimum values are 0 scores, the maximum values are 3, higher scores mean a worse outcome ) on renal interstitial capillary biopsy as determined by light microscopy.
Phase 2: The changes from the baseline of cardiac function | 6 months
  The change of LVMI (left ventricular mass index，g/m^2) from the baseline
Phase 2: The changes from the baseline of pain | 6 months
  The scores changes of BPI (The Brief Pain Inventory, short form) from the baseline, each iteam is scored on a 0-10 scale, with higher scores indicating greater severity.
Phase 2: The changes from the baseline of gastrointestinal function | 6 months
  The scores changes of GSRS (Gastrointestinal Symptom Rating Scale) from the baseline the minimum values are 0 scores, the maximum values are 35, higher scores mean a worse outcome

SECONDARY OUTCOMES:
eGFR | 52 weeks
  eGFR change from baseline in mL/min/(1.73m^2)
Cardiac function | 52 weeks
  LVMI change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, Principal Investigator — The General Hospital of Eastern Theater Command
Locations (3):
- China (3):
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
All data will be generated in this study are the property of Hangzhou Jiayin and should be kept strictly confidential together with the information provided by Hangzhou Jiayin. Investigator or any other delegated staff are not permitted to independently analyze and/or publish these data without the prior written authorization of Hangzhou Jiain.